CLINICAL TRIAL: NCT04694339
Title: Minority Barriers to Professional Advancement in Anesthesia
Brief Title: Minority Barriers in Anesthesia
Status: Recruiting | Type: Observational
Sponsor: Tufts Medical Center (Other)
Collaborators: American Society of Anesthesiologists (Other)
Responsible Party: Sponsor
Other Study IDs: STUDY00001139
Record Dates: First submitted 2021-01-02; First posted 2021-01-05 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Minority Barrier; Lack of Mentoring Program; Pass Over for Promotion
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Survey — Survey

SUMMARY:
The investigators aim to survey members of the ASA (medical students, residents, and attendings) who self-identify as minorities to assess if there are systemic barriers to minorities pursuing leadership positions. The investigators hypothesize that structural issues such as a lack of formalized mentoring programs play a role in reduced minority professional advancement.

DETAILED DESCRIPTION:
Within the American Society of Anesthesiology (ASA) underrepresented minorities comprise only 6.0% of leadership. Within the ASA, women additionally only hold 21% of House of Delegates and state society officer positions, while comprising 38% of the national anesthesiology workforce.

The investigators will be using a survey via SurveyMonkey with potential for an opt-in phone or Zoom interview via the interviewee using the contact information at the bottom of the SurveyMonkey. The questions for the Survey Monkey are below. The investigators will use the Tufts HIPAA-compliant Zoom account for any Zoom interviews.

In order to deidentify the phone and Zoom interviews, investigators will not label any transcripts of the interviews with names or identifying information. The investigators will also destroy all correspondence after a time and date for the phone/Zoom interview is set.

Participants will be self-selecting for this survey. The investigators aim to email the coordinators of the ASA (medical student component, resident component, general body) who will then forward investigators' contact letter and survey to participants' constituents. Given the self-selecting nature of the survey, the investigators are not specifically targeting individuals who identify as minorities--as there are variable definitions to this term--but rather investigators will use the survey to evaluate for trends within the responses. The investigators hypothesize that gender/race/sexual orientation may play a role in career choices for individuals, which will be elucidated through the survey responses. The investigators will sort the surveys into groups to where minority identification played a large role in career versus where it did not and then calculate the trend as a percentage of the total survey responses.

The investigators recognize that it may be more possible to provide in-depth responses to the survey via a phone or Zoom interview. Therefore, investigators have included a contact information in the contact letter and the Survey Monkey and will give participants the option of doing a phone/Zoom interview instead of the Survey Monkey.

Survey Questions:

Why did you decide to pursue medicine as a career? Why anesthesia? Did gender play a role in your decision to pursue medicine? In your decision to do anesthesia? Did race play a role in your decision to pursue medicine? In your decision to do anesthesia? Do you have any regrets about your career choice? Where do you currently practice? What led you to choose that practice setting? What mentorship resources were available to you along your career path? What is a professional success you had? What is a perceived failure you may have had? How did that effect your career? What if your five-year plan? Ten-year plan? Twenty? What is a minority?

ELIGIBILITY:
Inclusion Criteria:

* Members of ASA, medical students, residents, attending anesthesiologists, self-identifying as minorities

Exclusion Criteria:

* Non-ASA members

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Medical students, residents, attending anesthesiologists, members of ASA, self-identifying as minorities
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2020-12-22 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Minority barriers | through study completion, an average of 6 months
  The goal of this study is to highlight systemic barriers to minority advancement in anesthesia (Passed for promotion, lack of pay raises, lack of mentoring programs, how many times it happened during carrier). Responses will be reported as percentages, higher values mean barriers are more prevalent

CONTACTS AND LOCATIONS:
Overall Officials: Shara S Azad, MD, Study Director — Tufts Medical Center; Neeti Sadana, MD, Principal Investigator — Tufts Medical Center
Locations (1):
- Iwona Bonney, Boston, Massachusetts, United States